CLINICAL TRIAL: NCT06978257
Title: Protocol of a Two-Arm Randomized Controlled Trial (RCT) of Digital Positive Affect Intervention Study
Brief Title: Digital Positive Affect Intervention Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Nur Hani Zainal, Presidential Young Professorship (PYP) Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUS-IRB-2024-877
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Mild to Moderate Anxiety and Depression
Keywords: anxiety; depression
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital positive affect intervention (PAI) (Experimental): Access to weekly evidence-based positive affect intervention delivered online via Qualtrics surveys, and access to thrice daily evidence-based prompts and ecological momentary assessments (EMAs) delivered via a mental health (MH) mobile application for the 6-week treatment period.
  Interventions: Behavioral: Digital positive affect intervention (PAI)
- Self-monitoring intervention (Active Comparator): Access to thrice-daily self-monitoring prompts and ecological momentary assessments (EMAs) delivered via a mental health (MH) mobile application for the 6-week treatment period.
  Interventions: Behavioral: Self-monitoring intervention

INTERVENTIONS:
Behavioral: Digital positive affect intervention (PAI) — The Positive Affect Intervention (PAI) is a fully digital, self-guided program uniquely designed to deliver weekly 30-minute online sessions focused on cultivating positive emotions, meaning, and engagement, alongside daily ecological momentary prompts delivered thrice daily over six weeks. Distinctively, the intervention seamlessly integrates multimedia content (e.g., brief weekly videos introducing each session's core principles), practical exercises, and in-the-moment reflection, aiming to reinforce positive affect skills in real time. Its structure not only emphasizes proactive skill application through digital reminders but also systematically assesses user engagement and perceived helpfulness via ecological momentary assessments and post-session feedback questionnaires.
  Unlike conventional digital interventions that primarily focus on symptom reduction through passive content consumption, this PAI leverages continuous ecological momentary engagement via a dedicated mobile app, e
  Arms: Digital positive affect intervention (PAI)
Behavioral: Self-monitoring intervention — The self-monitoring intervention serves as an active comparator designed to isolate the effects of mood self-awareness without introducing therapeutic content. Participants in this arm receive daily prompts via the Qualtrics mEMA mobile app, three times per day over a six-week period, instructing them to track their mood and emotional states through brief ecological momentary assessments (EMAs). Unlike the digital positive affect intervention, this arm does not include psychoeducational material, skills training, or active enhancement strategies; instead, it focuses solely on routine self-monitoring to control for digital engagement and expectancy effects. This minimalist structure allows for a clean contrast between passive self-observation and active therapeutic engagement, enabling robust evaluation of the added value of the Positive Affect Intervention beyond self-monitoring alone
  Arms: Self-monitoring intervention

SUMMARY:
Anxiety and depression are highly prevalent mental health disorders that impose a significant burden on individuals and public health systems worldwide (GBD 2019 Mental Disorders Collaborators, 2022). Although many existing treatments focus on symptom reduction through targeting negative emotions, fewer interventions specifically enhance positive emotional experiences, despite growing evidence that low positive affect is a key feature of both anxiety and depression. Face-to-face psychologist-led positive affect therapy (PAT) is a promising intervention that aims to cultivate positive emotions, engagement, and meaning, potentially leading to greater improvements in emotional well-being than traditional approaches (Craske et al., 2019). However, empirical evaluations of digitally-delivered, asynchronously-coached, scalable versions of the PAT remain limited (Craske et al., 2024; Firth et al., 2017). The present study thus aims to investigate the comparative efficacy of a digital positive affect intervention (PAI) in reducing symptoms of anxiety and depression and enhancing overall mental health outcomes. We utilize a two-arm randomized controlled trial (RCT) design to investigate the effectiveness of a six-week digitally delivered positive affect intervention (vs. self-monitoring active control; Zainal & Newman, 2023) in reducing self-reported symptoms of anxiety and depression, as well as other secondary psychosocial outcomes, including sleep quality, quality of life, and emotion regulation. The treatment program comprises weekly evidence-based therapeutic material delivered online, and daily mental health (MH) mobile application prompts delivered thrice a day for the 6-week treatment period, based on evidence-based positive affect therapy principles. The active comparator comprises self-monitoring MH mobile application prompts for the 6-week treatment period. All participants will be assessed on several psychosocial outcomes at mid-treatment, post-treatment, and at 3-, 6-, and 12-month follow-up. The study hypothesizes that participants randomized to the digital PAI will experience greater improvement in anxious and depressive symptoms both immediately after treatment and up to a year later, compared to the self-monitoring MH app. Findings will contribute to growing evidence that digital PAI is an efficacious and feasible treatment to target and enhance positive emotions and related mental health outcomes in adults experiencing anxiety and depression.

DETAILED DESCRIPTION:
The present two-arm randomized controlled trial rigorously evaluates the efficacy of a six-week digitally-delivered positive affect intervention (PAI) compared to a self-monitoring active control among adults reporting symptoms of anxiety or depression. Participants (N=2400), recruited from the National University of Singapore and the broader community, are randomized to one of two arms: (1) the PAI, which provides weekly evidence-based therapeutic content via Qualtrics alongside daily ecological momentary prompts via mEMA Ilumivu platform to cultivate positive affect, or (2) an active control that engages participants in mood self-monitoring through a mental health mobile application. The intervention is designed to target positive emotion enhancement as a core mechanism for improving emotional well-being, reducing anxious and depressive symptoms, and bolstering resilience factors. Assessments are administered at baseline, mid-intervention (Week 3), post-intervention (Week 6), and follow-ups at 3, 6, and 12 months, capturing a comprehensive suite of psychosocial outcomes including quality of life, sleep quality, and emotion regulation capacities.

The study further investigates mediators and moderators to elucidate how and for whom the intervention confers benefit, providing granular insight into mechanisms of change. Subjects in the PAI arm also complete post-treatment assessments of satisfaction and cultural relevance to assess acceptability and contextual fit, an important consideration for digital mental health interventions (DMHIs). Both arms receive regular ecological momentary assessments three times daily to reinforce engagement and capture in-the-moment affective experiences. With its fully digital, scalable design, the trial not only tests clinical effectiveness but also addresses feasibility and user engagement, contributing meaningfully to the growing literature on positive emotion-focused digital interventions and their potential for integration into stepped-care mental health frameworks. This work is poised to advance understanding of digital therapeutic strategies that extend beyond symptom reduction to actively build psychological resilience and flourishing.

ELIGIBILITY:
Inclusion criteria

* Adults aged between 21 and 64 years
* Proficient in written and spoken English
* Ability to provide informed consent
* Scores between 5 and 14 on the Generalized Anxiety Disorder-7 (GAD-7) scale OR
* Scores between 5 and 19 on the Patient Health Questionnaire-9 (PHQ-9) scale
* Scores below 6 on the Altman Self-Rating Mania (ASRM) scale
* Possess an active smartphone with a valid Singapore phone number
* Mainly based in Singapore, within the next 15 months Exclusion criteria
* Failure to meet the above inclusion criteria
* Significant suicidal thoughts within the past two weeks, defined as self-reporting "more than half the days" or "nearly every day" on the PHQ-9 Item 9.
* Received psychiatric diagnoses of bipolar disorder, disorders of psychosis, severe clinical anxiety, or severe clinical depression.
* Severe clinical anxiety (scores of 15 to 21 on the GAD-7)
* Severe clinical depression (scores of 20-27 on the PHQ-9)

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Generalized Anxiety Disorder Symptoms at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  Generalized Anxiety Disorder-7 (GAD-7) scale contains 8 items measuring the frequency and intensity of anxiety symptoms, rated on a scale of 0-3 (0 = not at all, 3 = nearly every day). Higher scores reflect a greater reduction in anxiety symptoms.
Change from baseline Generalized Anxiety Disorder symptoms at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  Generalized Anxiety Disorder-7 (GAD-7) scale contains 8 items measuring the frequency and intensity of anxiety symptoms, rated on a scale of 0-3 (0 = not at all, 3 = nearly every day). Higher scores reflect a greater reduction in anxiety symptoms.
Change from baseline depressive symptoms at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  Patient Health Questionnaire-9 (PHQ-9) measures the severity and frequency of depressive symptoms with nine items rated on a scale of 0 to 3 (0 = not at all, 3 = nearly every day). Higher scores indicate a greater reduction in depressive symptoms.
Change from baseline depressive symptoms at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  Patient Health Questionnaire-9 (PHQ-9) measures the severity and frequency of depressive symptoms with nine items rated on a scale of 0 to 3 (0 = not at all, 3 = nearly every day). Higher scores indicate a greater reduction in depressive symptoms.

SECONDARY OUTCOMES:
Change from baseline emotion regulation strategies at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  The Emotion Regulation Questionnaire (ERQ) measures individuals' tendencies to regulate their emotions through cognitive reappraisal and expressive suppression. 10 items are rated on a scale of 1 to 7 (1 = strongly disagree, 7 = strongly agree). Higher scores indicate higher tendency to use that particular emotion regulation strategy.
Change from baseline emotion regulation strategies at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Emotion Regulation Questionnaire (ERQ) measures individuals' tendencies to regulate their emotions through cognitive reappraisal and expressive suppression. 10 items are rated on a scale of 1 to 7 (1 = strongly disagree, 7 = strongly agree). Higher scores indicate higher tendency to use that particular emotion regulation strategy.
Change from baseline automatic thoughts at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  The Automatic Thoughts Questionnaire (ATQ) assesses the frequency of negative automatic thoughts associated with depression. Eight items are rated on a scale of 1 to 5 (1 = not at all, 5 = all the time). Higher scores indicate greater reductions in the frequency of negative thoughts.
Change from baseline automatic thoughts at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Automatic Thoughts Questionnaire (ATQ) assesses the frequency of negative automatic thoughts associated with depression. Eight items are rated on a scale of 1 to 5 (1 = not at all, 5 = all the time). Higher scores indicate greater reductions in the frequency of negative thoughts.
Change from baseline attentional control at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  The Attentional Control Scale (ACS) assesses individuals' ability to focus and shift attention in the presence of distractions. 20 items are rated on a scale of 1 to 4 (1 = almost never, 4 = always). Higher scores indicate greater reductions in problems with regulating attention efficiently.
Change from baseline attentional control at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Attentional Control Scale (ACS) assesses individuals' ability to focus and shift attention in the presence of distractions. 20 items are rated on a scale of 1 to 4 (1 = almost never, 4 = always). Higher scores indicate greater reductions in problems with regulating attention efficiently.
Change from baseline self-compassion at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  The Self-Compassion Scale - Short Form (SCS-SF) assesses the frequency of self-compassionate behaviors and provides an evaluation of how individuals treat themselves during difficult times. 12 items are rated on a scale of 1 to 5 (1 = almost never, 5 = almost always). Higher scores indicate greater increases in self-compassion.
Change from baseline self-compassion at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Self-Compassion Scale - Short Form (SCS-SF) assesses the frequency of self-compassionate behaviors and provides an evaluation of how individuals treat themselves during difficult times. 12 items are rated on a scale of 1 to 5 (1 = almost never, 5 = almost always). Higher scores indicate greater increases in self-compassion.
Change from baseline mental well-being at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  The Mental Health Continuum - Short Form (MHC-SF) assesses overall mental well-being across emotional, psychological, and social dimensions. 17 items are rated on a scale of 0 to 5 (0 = never, 5 = every day). Higher scores indicate greater increases in flourishing.
Change from baseline mental well-being at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Mental Health Continuum - Short Form (MHC-SF) assesses overall mental well-being across emotional, psychological, and social dimensions. 17 items are rated on a scale of 0 to 5 (0 = never, 5 = every day). Higher scores indicate flourishing.
Change from baseline positive affect at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  The Positive and Negative Affect Schedule (PANAS) - PA subscale measures the extent to which an individual experiences positive emotion. 10 items are rated on a scale of 1 to 5 (1 = very slightly or not at all, 5 = extremely). Higher scores indicate greater increases in positive affect.
Change from baseline positive affect at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Positive and Negative Affect Schedule (PANAS) - PA subscale measures the extent to which an individual experiences positive emotion. 10 items are rated on a scale of 1 to 5 (1 = very slightly or not at all, 5 = extremely). Higher scores indicate greater increases in positive affect.
Change from baseline negative affect at 6 weeks post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Positive and Negative Affect Schedule (PANAS) - NA subscale measures the extent to which an individual experiences positive emotion. 10 items are rated on a scale of 1 to 5 (1 = very slightly or not at all, 5 = extremely). Higher scores indicate greater increases in negative affect.
Change from baseline negative affect at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Positive and Negative Affect Schedule (PANAS) - NA subscale measures the extent to which an individual experiences positive emotion. 10 items are rated on a scale of 1 to 5 (1 = very slightly or not at all, 5 = extremely). Higher scores indicate greater increases in negative affect.
Change from baseline anhedonia at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  The Dimensional Anhedonia Rating Scale (DARS) measures anhedonia by assessing desire, motivation, effort, and consummatory pleasure across four domains: hobbies, food/drink, social activities, and sensory experiences.17 items are rated on a 5-point scale of not at all to very much. Higher scores indicate greater reductions in anhedonia.
Change from baseline anhedonia at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Dimensional Anhedonia Rating Scale (DARS) measures anhedonia by assessing desire, motivation, effort, and consummatory pleasure across four domains: hobbies, food/drink, social activities, and sensory experiences.17 items are rated on a 5-point scale of not at all to very much. Higher scores indicate greater reductions in anhedonia.
Change from baseline positive valence at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  The Positive Valence Systems Scale (PVSS) assesses the positive valence system on several dimensions of rewards, food, physical touch and social interactions. Twenty-one items are rated on a scale of 1 to 9 (1 = extremely untrue of me, 9 = extremely true of me). Higher scores indicate stronger or more frequent responsiveness to a wide range of rewarding experiences.
Change from baseline positive valence systems at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Positive Valence Systems Scale (PVSS) assesses the positive valence system on several dimensions of rewards, food, physical touch and social interactions. 21 items are rated on a scale of 1 to 9 (1 = extremely untrue of me, 9 = extremely true of me). Higher scores indicate stronger or more frequent responsiveness to a wide range of rewarding experiences.
Change from baseline perceived stress at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  The Perceived Stress Scale (PSS) measures the degree to which individuals appraise situations in their lives as stressful, unpredictable, and uncontrollable. 10 items are rated on a scale of 0 to 4 (0 = never, 4 = very often). Higher scores indicate greater reductions in levels of perceived stress.
Change from baseline perceived stress at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Perceived Stress Scale (PSS) measures the degree to which individuals appraise situations in their lives as stressful, unpredictable, and uncontrollable. 10 items are rated on a scale of 0 to 4 (0 = never, 4 = very often). Higher scores indicate greater reductions in levels of perceived stress.
Change from baseline sleep quality at 6 weeks post-randomization | Baseline to 6 weeks post-randomization
  The Pittsburgh Sleep Quality Indicator (PSQI) assesses quality of sleep over a one-month period. The PSQI consists of 19 items that generate scores for seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. These components are summed to yield a global score ranging from 0 to 21. Higher scores indicate greater reductions in poor sleep quality.
Change from baseline sleep quality at 3, 6, and 12 months post-randomization | Baseline to 3 months, 6 months, and 12 months post-randomization
  The Pittsburgh Sleep Quality Indicator (PSQI) assesses quality of sleep over a one-month period. The PSQI consists of 19 items that generate scores for seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. These components are summed to yield a global score ranging from 0 to 21. Higher scores indicate greater reductions in poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore (NUS), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
At present, we are undecided about sharing individual participant data (IPD) because data governance, privacy considerations, and long-term storage protocols are still under review to ensure full compliance with institutional and regulatory guidelines. While we recognize the importance of data sharing for advancing scientific transparency and collaboration, any future decision to share IPD will be contingent on securing appropriate ethical approvals, ensuring participant confidentiality, and establishing secure data-sharing agreements that meet stringent data protection standards.

REFERENCES:
- [Background] Zainal NH, Newman MG. A randomized controlled trial of a 14-day mindfulness ecological momentary intervention (MEMI) for generalized anxiety disorder. Eur Psychiatry. 2023 Jan 16;66(1):e12. doi: 10.1192/j.eurpsy.2023.2. PMID 36645098
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Rizvi SJ, Quilty LC, Sproule BA, Cyriac A, Michael Bagby R, Kennedy SH. Development and validation of the Dimensional Anhedonia Rating Scale (DARS) in a community sample and individuals with major depression. Psychiatry Res. 2015 Sep 30;229(1-2):109-19. doi: 10.1016/j.psychres.2015.07.062. Epub 2015 Jul 26. PMID 26250147
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Khazanov GK, Xu C, Dunn BD, Cohen ZD, DeRubeis RJ, Hollon SD. Distress and anhedonia as predictors of depression treatment outcome: A secondary analysis of a randomized clinical trial. Behav Res Ther. 2020 Feb;125:103507. doi: 10.1016/j.brat.2019.103507. Epub 2019 Oct 31. PMID 31896529
- [Background] Keyes CL. The mental health continuum: from languishing to flourishing in life. J Health Soc Behav. 2002 Jun;43(2):207-22. PMID 12096700
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] GBD 2019 Mental Disorders Collaborators. Global, regional, and national burden of 12 mental disorders in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Psychiatry. 2022 Feb;9(2):137-150. doi: 10.1016/S2215-0366(21)00395-3. Epub 2022 Jan 10. PMID 35026139
- [Background] Firth J, Torous J, Nicholas J, Carney R, Pratap A, Rosenbaum S, Sarris J. The efficacy of smartphone-based mental health interventions for depressive symptoms: a meta-analysis of randomized controlled trials. World Psychiatry. 2017 Oct;16(3):287-298. doi: 10.1002/wps.20472. PMID 28941113
- [Background] Derryberry D, Reed MA. Anxiety-related attentional biases and their regulation by attentional control. J Abnorm Psychol. 2002 May;111(2):225-36. doi: 10.1037//0021-843x.111.2.225. PMID 12003445
- [Background] Craske MG, Meuret AE, Ritz T, Treanor M, Dour H, Rosenfield D. Positive affect treatment for depression and anxiety: A randomized clinical trial for a core feature of anhedonia. J Consult Clin Psychol. 2019 May;87(5):457-471. doi: 10.1037/ccp0000396. PMID 30998048
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- See also: Craske, M. G., Dunn, B. D., Meuret, A. E., Rizvi, S. J., & Taylor, C. T. (2024). Positive affect and reward processing in the treatment of depression, anxiety and trauma. Nature Reviews Psychology, 3(10), 665-685. https://doi.org/10.1038/s44159-024-00355 — https://doi.org/10.1038/s44159-024-00355-4
- See also: Hollon, S. D., & Kendall, P. C. (1980). Cognitive self-statements in depression: development of an automatic thoughts questionnaire. Cognitive Therapy and Research, 4, 383-395. https://doi.org/10.1007/bf01178214 — https://doi.org/10.1007/bf01178214